CLINICAL TRIAL: NCT00321048
Title: Spect Analysis of Cardiac Perfusion Changes After Whole Breast/Chest Wall Radiation Therapy With Active Breathing Coordinator
Brief Title: Spect Analysis of Cardiac Perfusion Changes After Whole Breast/Chest Wall Radiation Therapy With ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0609; NA_00002394 (Other: JHM IRB)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms; Carcinoma, Ductal; Adenocarcinoma
Keywords: breast cancer; SPECT; ABC device; Invasive adenocarcinoma of the left breast; Ductal Carcinoma In Situ of the left breast
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Left breast/chest wall irradiation with or without ABC (active breathing coordinator)

ARMS (2):
- ABC (Active Breathing coordinator) (Experimental): Patients are randomized to ABC arm will receive radiation with ABC. Cardiac perfusion will be assessed at baseline and 6 months after treatment and the difference will be compared to that seen in the No ABC arm.
  Interventions: Device: Active Breathing Coordinator
- No Active Breathing Coordinator (No Intervention): Patients randomized to the No ABC arm will receive radiation without ABC.Cardiac perfusion will be assessed at baseline and 6 months after treatment and the difference will be compared to that seen in the ABC arm.

INTERVENTIONS:
Device: Active Breathing Coordinator — A SPECT scan will be used to determine if the active breathing device reduces radiation toxicities.
  Arms: ABC (Active Breathing coordinator)

SUMMARY:
Cardiac perfusion changes have been seen after whole breast / chest wall irradiation for breast cancer. The Active Breathing Coordinator (ABC) device theoretically decreases radiation exposure to the heart during radiation for breast cancer. In this trial cardiac perfusion changes or lack thereof will be quantified in women treated with radiation for breast cancer while using the ABC device. The control group of the study will consist of patients randomized to radiation therapy without the ABC device.

DETAILED DESCRIPTION:
50 left sided breast cancer patients will be randomized to receive breast/chest wall irradiation with or without ABC. Patients will receive radiation therapy at a dose of 180-200 cGy per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed or mastectomy scar is at the discretion of the treating physician. The total dose to the tumor bed or mastectomy scar cannot exceed 6600cGy. Treatments will be given Monday through Friday.

After the completion of radiation therapy, patients will be seen on the following schedule:

A follow up examination will take place every 3-6 months for the first two years, then every 4-6 months for years for the next 3 years. After 5 years follow-up evaluations will occur annually. A SPECT scan will be obtained at 6 months post therapy.

Patients must be 18 and older and must have histologically confirmed (by routine H&E staining) invasive adenocarcinoma or Ductal Carcinoma In Situ of the left breast.

Patients must have also undergone a segmental mastectomy (SM) or Mastectomy.

Patients must not have received prior radiation therapy to the breast at any time for any reason.

Patients must not be pregnant due to the potential for fetal harm as a result of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 and older
* Patients must have histologically confirmed (by routine H&E staining) invasive adenocarcinoma or Ductal Carcinoma In Situ of the left breast.
* Patients must have undergone a segmental mastectomy (SM) or Mastectomy
* Patients must not have received prior radiation therapy to the breast at any time for any reason.
* Any patient with active local-regional disease prior to registration is not eligible.
* Patients must not be pregnant due to the potential for fetal harm as a result of this treatment regimen. Women of child-bearing age will be given a serum pregnancy test prior to study entry to ensure they are not pregnant. Women of child-bearing potential must use effective non-hormonal contraception while undergoing radiation therapy.
* Patients must not have a serious medical or psychiatric illness which prevents informed consent or compliance with treatment.
* All patients must be informed of the investigational nature of this study and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients requiring oxygen
* Sarcoma or Squamous Cell pathology
* Right-sided breast cancers
* Metastatic disease to the breast

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zellars, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center- Dept. Radiation Oncology
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zellars R, Bravo PE, Tryggestad E, Hopfer K, Myers L, Tahari A, Asrari F, Ziessman H, Garrett-Mayer E. SPECT analysis of cardiac perfusion changes after whole-breast/chest wall radiation therapy with or without active breathing coordinator: results of a randomized phase 3 trial. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):778-85. doi: 10.1016/j.ijrobp.2013.12.035. PMID 24606847

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Breathing Coordination: Patients will receive radiation therapy at a dose of 180-200 cGy per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed or mastectomy scar is at the discretion of the treating physician. The total dose to the tumor bed or mastectomy scar cannot exceed 6600cGy. Treatments will be given Monday through Friday.
  Patients in this group were treated with Active Breathing Coordinator:
  A SPECT scan will be obtained at baseline and at 6 months follow to determine changes in cardiac perfusion
- No Active Breathing Coordination: Patients will receive radiation therapy at a dose of 180-200 cGy per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed or mastectomy scar is at the discretion of the treating physician. The total dose to the tumor bed or mastectomy scar cannot exceed 6600cGy. Treatments will be given Monday through Friday.
  (Patient ARE NOT treated with ABC) A SPECT scan will be obtained at baseline and at 6 months follow to determine changes in cardiac perfusion
Period: Overall Study
Arm/Group | Active Breathing Coordination | No Active Breathing Coordination
Started | 28 | 29
Completed | 22 | 21
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected for participants who completed study interventions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Breathing Coordination | No Active Breathing Coordination | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Full Range); unit: years] | 52.8 [20 to 86] | 58.7 [35 to 85] | 55.8 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Active Breathing Coordinator (ABC) Device as Determined by the Mean Apical Perfusion Score
Description: Efficacy of the ABC device in protecting the heart from radiation (XRT) damage in patients with L breast cancer is determined by the change in cardiac perfusion (mean apical perfusion score) as measured by SPECT between baseline and 6 month follow up. A score of 1 represents an equivocal or mild reduction in perfusion, 2 represents moderately reduced perfusion, 3 represents severely reduced perfusion, and 4 indicates absent perfusion.
Time Frame: Baseline (pre-radiation) to 6 months (post-radiation)
Population: We understand the reporting score on a scale however, in this case the Mean Perfusion Score was utilized.
Measure: Mean (Standard Deviation); unit: Mean Perfusion Score
Arm/Group | Active Breathing Coordination | No Active Breathing Coordination
Number analyzed (Participants) | 22 | 21
Mean Perfusion Score
  Mean Apical Perfusion Pre XRT | 1.2 (0.9) | 2.0 (1.5)
  Mean Apical Perfusion Post XRT | 2.1 (1.5) | 2.5 (1.6)

ADVERSE EVENTS:
Time Frame: Baseline (pretreatment) to 48 months posttreatment)
Arm/Group | Active Breathing Coordination | No Active Breathing Coordination
All-Cause Mortality (participants affected / at risk) | 2/22 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No